CLINICAL TRIAL: NCT06018168
Title: A Randomized, Controlled Study Evaluating the Efficacy of a Skincare Routine and Acne Supplement or a Skincare Routine Alone on Improving Acne and Other Symptoms of PMS
Brief Title: An RCT Evaluating the Efficacy of a Skincare Routine and Acne Supplement on Improving Acne and Other Symptoms of PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clearstem Skincare (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20282
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Acne; Premenstrual Syndrome
MeSH Terms: conditions — Acne Vulgaris; Premenstrual Syndrome

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a randomized, controlled trial in which participants will be split into two groups. Both will use the skincare routine, but one group will also take the MINDBODYSKIN supplement in combination with the skincare routine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group One: Skincare Routine Only (Active Comparator): Participants will follow instructions for the skincare routine only. Participants will complete the routine twice daily.
  Interventions: Other: Skincare Routine
- Group Two: Skincare Routine + Supplement (Active Comparator): Participants will follow instructions for the skincare routine AND will take a daily supplement.
  Interventions: Other: Skincare Routine; Dietary Supplement: MINDBODYSKIN Supplement

INTERVENTIONS:
Other: Skincare Routine — Morning:
  1. GENTLECLEAN - Wash with a quarter-sized amount of lukewarm water. Pat skin dry after.
  2 CELLRENEW - Shake well, apply 2-3 pumps over the entire face, and massage into the skin 3. YOUARESUNSHINE - Apply generously and evenly as the last step in the skincare routine (before makeup).
  Night:
  1. VITAMINSCRUB - Wet your face with lukewarm water & apply a quarter-sized amount to wet palms. Lather until foamy. Gently massage the scrub using circular motions for 5-10 seconds. Rinse with lukewarm water and pat dry.
  2. CLEARITY - Apply 2-3 pumps and massage into the skin avoiding the eye area. Let sit for 10-15 minutes. Do not wash off.
  3. CELLRENEW - Shake well, apply 2-3 pumps over the entire face, and massage into the skin
  4. HYDRAGLOW - Apply a dime-size amount of lotion and massage into the face
Dietary Supplement: MINDBODYSKIN Supplement — Participants will take 3 capsules daily with a meal. The MINDBODYSKIN acne supplement contains Vitamin A (6,100mcg per serving of 3 capsules), Vitamin B12, Vitamin B-5, 5-Hydroxytryptophan (5-HTP), 3,3'-Diindolymethane (DIM), a proprietary liver blend of milk thistle, dandelion extract and L-glutathione, turmeric root extract, a proprietary digestive blend of protease and betaine hydrochloride, and silicon dioxide.
  Arms: Group Two: Skincare Routine + Supplement

SUMMARY:
This study aims to evaluate the efficacy of the MINDBODYSKIN Hormonal Acne Supplement and a prescribed skincare routine of 6 products on facial acne and on symptoms of PMS, compared to a skincare routine of 6 products alone. This study will last for 24 weeks. The study will be conducted as a randomized, controlled trial in which participants will be split into two groups. Both will use the skincare routine, but one group will also take the MINDBODYSKIN supplement in combination with the skincare routine.

ELIGIBILITY:
Inclusion Criteria:

Female 18 years of age or older Have regular acne Have any noticeable PMS symptoms like stress, bloating, mood swings, acne Be generally healthy (i.e. don't live with any uncontrolled chronic disease besides acne).

Have a body weight of >120 lbs.

Exclusion Criteria:

Have any pre-existing conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.

Be currently using any prescribed medications for their face Anyone with any known severe allergic reactions Women who are pregnant, breastfeeding or attempting to become pregnant Anyone unwilling to follow the study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Changes in facial acne. [Baseline to Week 24] | 24 weeks
  Participants will provide photos of their face for virtual skin grading by dermatologist.
Changes in blood serum levels of vitamin A. [Baseline to Week 24] | 24 weeks
  Participants will undergo blood draws to assess blood serum levels of vitamin A.
Changes in participants perception of facial acne. [Baseline to Week 24] | 24 weeks
  Survey-based assessment (0-5 scale) of participants perception of changes to their facial acne.

SECONDARY OUTCOMES:
Changes in symptoms of premenstrual syndrome (PMS). [Baseline to Week 24] | 24 weeks
  Survey-based assessment (0-5 scale) of common symptoms associated with PMS.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided